CLINICAL TRIAL: NCT01068821
Title: Randomized Controlled Trial Comparing Commonly Used Techniques to Prevent Slippage During Steep Trendelenburg's Position
Brief Title: Trendelenburg's Slide Prevention Study
Acronym: SPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mary Ellen Wechter, Independent Physician, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 09-000685-01
Record Dates: First submitted 2010-02-12; First posted 2010-02-15 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-04

CONDITIONS: Misadventure During Surgical Operation; Postoperative Complications
Keywords: Slide; Trendelenburg's position; Postoperative; neurologic complaints
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Egg crate foam mattress (Active Comparator): Patients will be placed on egg-crate foam mattress instead of a gel pad by randomization. All other positioning and measurements, including outcomes measures will be the same as for the the primary experimental intervention (gel pad).
  Interventions: Other: Egg crate foam mattress
- Gel pad (Active Comparator): Patients will be placed on gel pad instead of egg-crate foam mattress by randomization. All other positioning and measurements, including outcomes measures will be the same as for the the primary experimental intervention (gel pad).
  Interventions: Other: Gel pad

INTERVENTIONS:
Other: Gel pad — A gel pad (mattress) (approximately 3cm thick) is placed under the patient on top of the usual operating room mattress, directly in contact with patient's skin from buttocks to shoulders with the patient in dorsal lithotomy position under general anesthesia. Time in Trendelenburg's position and time operating are both recorded. The position of two bony landmarks (left anterior superior iliac spine and left acromioclavicular joint) are marked before Trendelenburg's position (30 to 45 degrees below horizontal) and immediately after returning the patient to horizontal position.
  Other Names: Gel Pad:; Allen Medical
  Arms: Gel pad
Other: Egg crate foam mattress — An egg-crate foam mattress (approximately 5cm thick) is placed under the patient on top of the usual operating room mattress, directly in contact with patient's skin from buttocks to shoulders with the patient in dorsal lithotomy position under general anesthesia. Time in Trendelenburg's position and time operating are both recorded. The position of two bony landmarks (left anterior superior iliac spine and left acromioclavicular joint) are marked before Trendelenburg's position (30 to 45 degrees below horizontal) and immediately after returning the patient to horizontal position.
  Other Names: Pink Foam:; Kendall Company, Ref# 31163457
  Arms: Egg crate foam mattress

SUMMARY:
The purpose of this study is to compare two cushioning materials (a gel mattress and an egg-crate foam mattress) placed beneath patients undergoing gynecologic surgery to prevent patients from sliding toward the head of the bed during head-down positioning.

Our hypothesis is that the two materials will be equally good at preventing slide on the table and that slide will be less than 5 cm (<2 inches) on average.

DETAILED DESCRIPTION:
Patient undergoing laparoscopic gynecologic surgery are often placed in steep (30 to 45 degrees) Trendelenburg's (head lower than feet) position. This helps the bowels to move towards the patient's head, making surgery in the pelvis safer. During surgery, if patients slide a great deal toward the head of the bed, nerve injury and hernia risk may be increased. Several techniques are in use to prevent patients from sliding on the bed during surgery, and of these, increasing the friction between a patient's skin and the bed surface appears to be the safest technique. Two materials are in use to increase this friction: a gel pad or an egg-crate foam mattress upon which the patient lies with bare skin. This study is comparing these two materials to see which material is associated with the LEAST amount of patient slide. Our hypothesis is that the two materials will be equally good at preventing slide on the table and that slide will be less than 5 cm (<2 inches) on average.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing gynecologic laparoscopic or robotic-assisted laparoscopic surgery
* Trendelenburg's position is planned
* General anesthesia is planned

Exclusion Criteria:

* Patients with intolerance of Trendelenburg's position
* Patients whose surgery are converted to laparotomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Wechter, MD, MPH, Principal Investigator — Mayo Clinic, Baptist Medical Center
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- [Background] Klauschie J, Wechter ME, Jacob K, Zanagnolo V, Montero R, Magrina J, Kho R. Use of anti-skid material and patient-positioning to prevent patient shifting during robotic-assisted gynecologic procedures. J Minim Invasive Gynecol. 2010 Jul-Aug;17(4):504-7. doi: 10.1016/j.jmig.2010.03.013. Epub 2010 May 14. PMID 20471916

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with planned laparoscopic or robotic procedures were offered participation in the preoperative holding area. Recruitment started 3/1/2010 and ended 5/10/2010.
Pre-assignment Details: Patients were enrolled if they acknowledged their desire to participate. Patients were excluded if they were brought to the operating room before being approached for participation or if they indicated they did not wish to participate. The materials being compared are already both commonly used for gynecologic surgery.
Groups:
- Gel Pad: Patients will be placed on gel mattress instead of egg-crate foam mattress by randomization. All other positioning and measurements, including outcomes measures will be the same as for the the primary experimental intervention (gel pad).
Period: Overall Study
Arm/Group | Egg Crate Foam Mattress | Gel Pad
Started | 31 | 29
Completed | 30 (1 patient had slide measured, but her patient ID not listed; couldn't do postoperative followup.) | 29
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Egg Crate Foam Mattress | Gel Pad | Total
Number analyzed (Participants) | 31 | 29 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 22 | 45
  >=65 years | 8 | 7 | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.8) | 53.6 (12.7) | 54.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 31 | 29 | 60

OUTCOME MEASURES:

1. Primary Outcome: Amount of Patient Movement on the Operating Room Table
Description: Patients undergoing gynecologic surgery require steep (30 to 45 degree) Trendelenberg's position to allow adequate exposure of the pelvis. This position leads to a small amount of movement toward the head of the bed. The table was marked at the point of the anterior superior iliac spine (ASIS) and at the point where a vertical marker touching the acromioclavicular (AC) joint of the left shoulder drops to the table. At the end of the surgery, when the operating table is leveled, the final positions of ASIS and AC will be measured. Measurements were made in centimeters to the tenth position.
Time Frame: About 150 minutes after start of surgery
Population: Study size calculation was performed for 80% power, and p=0.05
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Egg Crate Foam Mattress: Patient positioned on egg crate foam mattress during surgery
- Gel Pad: Patient positioned on gel pad during surgery
Arm/Group | Egg Crate Foam Mattress | Gel Pad
Number analyzed (Participants) | 30 | 29
centimeters | 3.2 (1.9) | 4.5 (4.0)
Statistical Analysis 1: Comparison: Egg Crate Foam Mattress vs Gel Pad; Sample size calculations (yielding 25 patients per group): two-sided 5% significance level and a power of 80% for detection of a 2 cm (SD 2.5 cm) difference. Continuous variables analyzed by Student's T-test and One way Analysis of Variance (ANOVA) with statistical significance: p value ≤ 0.05 or 95% Confidence Interval excluding one. Confirmation by Wilcoxon Rank-Sum/Mann-Whitney and Kruskal-Wallis tests. Categorical variables by Chi Square Test, confirmed by Fisher's Exact test; Test type: Superiority or Other; p = 0.1, t-test, 2 sided

2. Secondary Outcome: Number of Participants Reporting a Neurologic Deficit in Extremities After Surgery
Description: The neurologic deficit was assessed as follows: Patients' postoperative care was unchanged from routine for this study. Any postoperative complaints regarding limb pain or weakness or numbness were recorded and assessed with neurologic exam to determine sensation or motor components. Absence of resolution was documented.
Time Frame: postoperative day 1 and postoperative week 3-8
Population: Participants were analyzed per protocol if they returned for postoperative followup (59 of 60 were analyzed)
Measure: Number; unit: participants
Arm/Group | Egg Crate Foam Mattress | Gel Pad
Number analyzed (Participants) | 30 | 29
participants | 0 (0) | 3 (0.19)
Statistical Analysis 1: Comparison: Egg Crate Foam Mattress vs Gel Pad; Fischer's exact test, significance defined as p<0.05; Test type: Superiority or Other; p = 0.5, Fisher Exact

ADVERSE EVENTS:
Time Frame: Participants were followed from randomization until final chart review at study end: Mean follow up surveillance of 344.9 days (SD 116.2)
Arm/Group | Egg Crate Foam Mattress | Gel Pad
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

LIMITATIONS AND CAVEATS:
Evaluation of postoperative outcomes was non-systematic using chart review for all participants except for one participant whose identity was not listed on data abstraction sheet.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No